CLINICAL TRIAL: NCT03537989
Title: Perioperative Fluid Treatment in Colorectal Surgery
Brief Title: Restricted Fluid Therapy in Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Glostrup University Hospital, Copenhagen (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other); Vejle Hospital (Other); Aalborg University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Brandstrup, Chief Surgeon, Clinical Associate Professor, PhD, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2018-05-11; First posted 2018-05-25 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Surgery; Postoperative Complications
Keywords: fluid therapy; Restricted fluid therapy; saline
MeSH Terms: conditions — Postoperative Complications | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restricted group (Experimental): Oral fluid to 2 h before surgery. Intra-operatively: Glucose 5% (500 ml - volume drunk during fast); HAES 6% for blood loss volume to volume; IV-medicine in saline 0.9% for anesthesia and antibiotics. Blood products after current rules.
  Postoperatively: 1000 ml glucose containing fluid in the recovery room. Free oral intake of fluid and food as well as enteral feeding by tube 500 ml.
  In the wards: Enteral feeding by tube 1000 ml postoperative day 1-3. Free fluid and food by mouth. If less than 1500 ml fluid pr. mouth supplement with VI-fluid.
  Pathological fluid loss (high output stoma, aspirate, vomit etc.) - replace with IV-fluid. Goal: zero fluid balance with up to 1-kilogram body weight increase.
  Urine < 0.5 ml/kg/h: supplement with fluid. MAP < 60 and hypovolemia: treat with fluid.
  Interventions: Drug: Saline
- Standard group (Active Comparator): Oral fluid to 2 h before surgery. Intra-operatively: Saline 500 ml for fasting; 500 ml HAES 6% for the epidural, Saline for the third space: 7 ml/kg/h first hour, 5 ml/kg/h 2.-3. Hour, 3 ml/kg/h subsequent hours. 1000-1500 ml Saline replaced lost blood up to 500 ml, additional HAES 6% for additional blood loss; IV-medicine in saline.
  Postoperatively: 1000-2000 ml isotonic fluid in the recovery room. Free oral fluid and food as well as enteral feeding by tube 500 ml.
  In the wards: Enteral feeding by tube 1000 ml postoperative day 1-3. Free fluid and food by mouth. Supplemental iv-fluid according to department rules. Pathological fluid loss (high output stoma, aspirate, vomit etc.) - replace with IV-fluid.
  Urine < 0.5 ml/kg/h: supplement with fluid. MAP < 60 and hypovolemia: treat with fluid.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — To reduce the volume of saline administered during surgery of the colon and the rectum
  Other Names: NaCl 0.9%

SUMMARY:
This is a protocol for a trial carried out from 1999 to 2002. At that time, surgical patients received a large volume of intravenous saline during operations on the colon or the rectum, often so much fluid that their bodyweight increased by 4-6 kilograms. We hypothesized; that a restricted fluid regimen could prevent the development of cardiopulmonary complications and improve wound healing including the healing of an anastomosis of the gut.

We designed a clinical randomized assessor blinded multi-center trial comparing a restricted fluid regimen to a standard fluid regimen, the difference being the volume of saline administered to the patients. Patients undergoing surgery on the colon or the rectum were included after informed oral and written consent.

The restricted regimen aimed at zero-fluid balance with allowance for a body weight increase of 1 kg. The standard regimen was a bit "dryer" than the actual standard; our patients in the standard group received saline causing a body weight increase of only 3-4 kg. The fluid therapy started at midnight the day of operation, went on through the operation and continued on the wards until discharge. The patients were encouraged to eat and drink as much and as soon as possible after the operation.

The primary outcome was the number of patients who died or suffered a complication measured within 30 days of surgery. We looked at all complications, but especially heart and lung complications and complications related to the healing of wounds and anastomosis.

The patients was examined in the outpatient clinic after 30 days, and in addition, blinded assessors were reviewing the medical files for registration of postoperative complications.

The results are published in The Annals of Surgery 2003; 238(5)641-48. The restricted regimen nearly halved the number of patients with complications, and heart and lung complications were almost eliminated.

Other investigators confirmed the results, and a more restricted approach to fluid therapy to surgical patients has been implemented worldwide.

DETAILED DESCRIPTION:
Aim:

To show the effect of a restrictive fluid regime compared to a standard regime by the frequency of complications in patients undergoing colorectal surgery.

Background:

Previous studies have risen suspicions of fluid balance, and especially a large amount of water and NaCl administration, can be a significant factor in developing postoperative complications (1, 2).

In 1990 in Critical Care Magazine, Lowell et al. described patients who in transferring to intensive therapy had an increased weight of > 10% of their preoperative weight, had a significantly higher mortality rate of 31.6 % than patients with an increased weight of < 10%, who only had a mortality rate of 10.3 %.

Some studies, have described, how all patients undergoing gastroenterological operations increase their body weight by 2-4% of the preoperative weight during the first 24 hours following surgery due to the perioperative saline intravenously (2, 3). The patients have been given a median of 6-7 L saline intravenously during the day of operation. This is fully comparable to other studies (3, 5).

Based on previous guidelines in anesthesiological departments, a volume of saline of 15 ml/kg bodyweight was administered during the first hour of surgery, and 7.5 ml/kg during the following hours. Furthermore, any blood loss was replaced by 2.5 ml saline per ml blood lost (6-9).

The patients in the study by Beier-Holgersen et al. returned to their preoperative weight after 4-5 days. In this material of 60 patients, six patients developed leakage of the bowel anastomosis, and two patients died from AMI and ARDS. Nine patients with severe complications had a weight gain of 6-14%.

The increased postoperative fluid retention results in increased universal edema, which can significantly affect the tissue's microcirculation and oxygenation. This may have influenced the healing of intestinal anastomoses and the development of cardiovascular and pulmonary complications, which typically occurred during the third postoperative day. Based on this, it is therefore relevant to investigate whether perioperative intervention against fluid administration can improve the postoperative course.

Design:

Prospective randomized multicenter study with stratification for each center. Block randomization with four patients per block. It is necessary to incorporate several centers for the investigation to be finished within a reasonable time.

Material:

Two x 70 patients scheduled for colorectal resection. The number is determined from previous works (1, 2) finding a total complication rate of at least 30% after colorectal resection in post-operatively early-nourished patients. The investigators wish to reduce this to 10% (MIREDIF = 20%). The risk of Type 1 error (5%) is set low to avoid overlooking a possible gain. The risk of Type 2 error is set at 20% (power at 80%).

As the material is unlikely to meet the normal distribution, the number of participant's increases to 70 in each group, i.e. 140 patients must be included. In order to reduce the variation, each center must include at least 16 patients (which means that up to nine centers have to participate).

Method:

1. Patients are included preoperatively after informed consent. An investigator at the local center randomize the patients to either standard fluid treatment or restrictive perioperative fluid treatment. The main difference between the two regimes is that less isotonic saline is administered in the restrictive regime. Anesthesia and postoperative nutrition regimes are the same in the two groups. The patients are ASA and Apache 2 scored.
2. Weight registration: The patient is weighed on the same set of scales at the time of hospitalization (entry weight), after bowel cleansing, and in the morning on the day of operation (preoperative weight). Hereafter daily weighing every postoperative morning.
3. Blood tests: Blood is withdrawn on the day of hospitalization, on the day of operation in the morning, on arrival in the recovery ward and the following 7 days (or until discharged).
4. Anesthesia: Patients must fast for food from midnight before surgery, but they can have clear fluids up to 2 hours preoperatively, but max. 500 ml from midnight.

   Premedication is a tablet of Triazolam 0.125 mg with 50-100 ml of water by mouth.

   Combined epidural and general anesthesia are used: An epidural catheter is inserted corresponding to TH10-12, tested with Lidocaine 2% and adrenaline 3-4 ml. After 3-5 minutes this is supplemented with refracted doses of Bupivacaine 0.5% until the blockade is sufficient (often about 8-12 ml). Continuous infusion of Bupivacain is administered 0.5%, 4-8 ml/hour. Finally, a bolus injection of 2 mg Morphine is administered. General anesthesia is induced with Fentanyl 5μg/kg, Thiopental 3-4 mg/kg and Rocuronium (Esmeron®) 0.6 mg/kg (all doses are modified according to each patient's needs and cardiovascular condition). Anesthesia is maintained with Isoflurane 0.2-0.4% end-tidal concentration in oxygen / atmospheric air (inspiratory oxygen concentration 30-35%). The neuromuscular block can be reverted with neostigmine when needed.

   Hypotension Diagnosis and Treatment: Detailed guidelines for clinical treatment and handling are given in the case report forms (CRF).
5. Perioperative fluid treatment: During operation, fluid is submitted and recorded in the CRF. Fluid balance is calculated at the end of anesthesia.
6. Monitoring: Standard anesthesia monitoring as recommended by Danish Anesthesiological Society. A central vein catheter (CVK) is placed if needed after the initiation of anesthesia to measure central venous pressure (CVP) until the patient is discharged from the recovery ward. Arterial blood gases and hematocrit are withdrawn immediately after the initiation of anesthesia, immediately after arriving at the recovery ward and before the patient is transferred to the surgical ward, in addition to clinical needs.
7. Surgery: Surgery is performed in accordance with the department's routines. During the surgery, a nutritional feeding tube is inserted in the duodenum for postoperative enteral nutrition. If the tube cause nausea, the tube is removed and the patient will consume nutrition according to ability by mouth.

   Antibiotic prophylaxis, bowel cleansing, physiotherapy, etc. follow the usual guidelines of the respective departments.
8. Postoperative fluid treatment and nutrition during the day of operation: Fluid recordings continue from the end of the anesthesia, on the recovery ward and for the rest of the day of operation. On the day of operation, 600 ml of Nutri-concentrated 75 is given in the feeding tube. Nutri-concentrated 75 contains 200 kcal and 7.5 g protein per 100 ml. 1000 ml pr. Day cover the recommended daily allowances for vitamins and minerals.
9. Fluid treatment and nutrition in the following days: Nutri-concentrated 75® 1000 ml/day is continued the first three postoperative days. Thereafter the patient is expected to eat normally. The fluid regime in the restrictive group assessed based on the patient's weight, ability to drink independently and blood samples. The standard regime follows the department's usual postoperative regime.
10. Postoperative analgesia: The basis is an epidural infusion of the standard mixture of Bupivacain-Morphine (5 mg Morphine + 250 mg Bupivacain in NaCl to the volume of 100 ml), 4-8 ml/hour. In addition, Morphine 5-10 mg p.n. If there are no contraindications, Paracetamol or NSAID can be administered (orally or rectally). The epidural pain treatment is continued postoperatively for a maximum of 4 days, after which the epidural catheter is removed. If the patient need analgesics hereafter, opioid is given by mouth or intravenously as well as Paracetamol and/or NSAIDs.
11. For the treatment of nausea the following may be given: Ondansetron (Zofran®), Cisapride (Prepulsid®), Metoclopramide (Primperan®) or DHB.
12. A postoperative outpatient visit with the investigating doctor is planned 4 weeks after the surgery. Postoperative complications are registered.

Ethics:

Participation in the project is voluntary and inclusion is after informed consent. Consent can be withdrawn at any time without further explanation, and without this affecting the patient's treatment in any way.

There is no risk associated with participation in the project, but discomfort associated with additional blood sampling for the project, no more than 4-5 times. However, these blood samples will preferably be taken from the CVK, so the patient avoids being stabbed unnecessarily.

In the long term, a treatment benefit is possible and this appears to outweigh the discomfort mentioned above.

The project is registered with the Scientific Ethics Committee (multicenter study) and The Danish Data registration agency in accordance with applicable guidelines. All person-identifiable data is destroyed after the project is completed.

Addendum to the protocol written during the patient inclusion and before the trial was completed.

Hypothesis:

Both too little and too much fluid administered intravenously may be harmful to the cardiac function (low oxygen supply and congestion) and cause cardiovascular complications: Postoperatively developed arrhythmias, AMI, pneumonia, pulmonary congestion, postoperatively developed pleural exudate, pulmonary edema or ARDS.

Both too little and too much fluid administered intravenously may be harmful to tissue healing (low oxygen supply and interstitial edema) and cause complications related to tissue healing and infection: Infections of the wound, bursting of the wound (superficial and deeper), leakage from the anastomosis and separation of stoma.

Randomization:

The investigating surgeon or anesthesiologist perform the randomization by opening consecutively numbered opaque envelopes. The randomization is stratified for each center and for colonic and rectal surgery the latter by opening an envelope with highest number for rectal surgical patients, and with lowest number for colonic patients.

Blinding:

Specialist surgeons reading the medical journals censored for all information about randomization group, fluid therapy given or bodyweight measurements will perform a blinded assessment for the primary outcome.

Two doctors will evaluate each patient file, and in case of disagreement, a third will decide the outcome.

Plan for analysis:

An intention to treat analysis will be performed for the primary outcome for all patients included in the trial whether or not they met a post randomization exclusion criterion, and therefore did or did not receive the allocated treatment.

A per protocol analysis will be performed for the primary outcome for all patients fulfilling the in- and exclusion criteria whether or not they adhered to the protocol.

Subgroup analysis will be performed for the patients with Major-, Minor-, Cardio-pulmonic- and tissue-healing complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for planned surgery on the colon or the rectum
* ASA group 1-3

Exclusion Criteria:

• Patients unable to give informed consent (mental disorders, dementia, language problems)

Patients with:

* Diabetes mellitus
* Renal insufficiency
* Disseminated cancers or secondary cancers
* Inflammatory bowel disease
* Diseases hindering epidural analgesia
* Alcohol consumption more than 35 drinks pr. Week
* Pregnant and lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 1999-11-01 (Actual); Primary Completion 2001-08-31 (Actual); Study Completion 2001-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications and mortality | After 30 days of follow-up
  The complications was defined by protocol.

SECONDARY OUTCOMES:
Cardiopulmonary complications | After 30 days of follow-up
  AMI, debut of cardiac arrhythmias, pulmonary congestion, pulmonary oedema, ARDS, pneumonia
Complications related to tissue healing | After 30 days of follow-up
  Wound complications and anastomotic leak

OTHER OUTCOMES:
Hospital stay | after 30 days of follow-up
  Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Brandstrup, PhD, Principal Investigator — Holbaek Hospital

IPD SHARING:
Plan to Share IPD: Undecided
We do not mind sharing the data

REFERENCES:
- [Background] Lowell JA, Schifferdecker C, Driscoll DF, Benotti PN, Bistrian BR. Postoperative fluid overload: not a benign problem. Crit Care Med. 1990 Jul;18(7):728-33. doi: 10.1097/00003246-199007000-00010. PMID 2364713
- [Background] Beier-Holgersen R, Boesby S. Influence of postoperative enteral nutrition on postsurgical infections. Gut. 1996 Dec;39(6):833-5. doi: 10.1136/gut.39.6.833. PMID 9038665
- [Background] Nielsen OM, Engell HC. Increased glomerular filtration rate in patients after reconstructive surgery on the abdominal aorta. Br J Surg. 1986 Jan;73(1):34-7. doi: 10.1002/bjs.1800730113. PMID 3947870
- [Background] Rasmussen LA, Rosenberg J, Crawford ME, Kehlet H. [Perioperative fluid therapy. A quality control study]. Ugeskr Laeger. 1996 Sep 16;158(38):5286-90. Danish. PMID 8966776
- [Background] Vamvakas EC, Carven JH, Hibberd PL. Blood transfusion and infection after colorectal cancer surgery. Transfusion. 1996 Nov-Dec;36(11-12):1000-8. doi: 10.1046/j.1537-2995.1996.36111297091746.x. PMID 8937412
- [Background] Cosnett JE. The origins of intravenous fluid therapy. Lancet. 1989 Apr 8;1(8641):768-71. doi: 10.1016/s0140-6736(89)92583-x. No abstract available. PMID 2564573
- [Background] Vermeulen LC Jr, Ratko TA, Erstad BL, Brecher ME, Matuszewski KA. A paradigm for consensus. The University Hospital Consortium guidelines for the use of albumin, nonprotein colloid, and crystalloid solutions. Arch Intern Med. 1995 Feb 27;155(4):373-9. doi: 10.1001/archinte.155.4.373. PMID 7848020
- [Background] Weinstein PD, Doerfler ME. Systemic complications of fluid resuscitation. Crit Care Clin. 1992 Apr;8(2):439-48. PMID 1568149
- [Result] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Derived] Brandstrup B, Beier-Holgersen R, Iversen LH, Starup CB, Wentzel LN, Lindorff-Larsen K, Petersen TC, Tonnesen H. The Influence of Perioperative Fluid Therapy on N-terminal-pro-brain Natriuretic Peptide and the Association With Heart and Lung Complications in Patients Undergoing Colorectal Surgery: Secondary Results of a Clinical Randomized Assessor-blinded Multicenter Trial. Ann Surg. 2020 Dec;272(6):941-949. doi: 10.1097/SLA.0000000000003724. PMID 31850996